CLINICAL TRIAL: NCT01924702
Title: Chronic Aphasia - Improved by Intensive Training and Electrical Brain Stimulation (CATS)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Charité Neurocure AG Flöel (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CATS02EO0801
Record Dates: First submitted 2013-08-14; First posted 2013-08-16 (Estimated); Last update posted 2015-02-04 (Estimated); Status verified 2015-02

CONDITIONS: Aphasia; Anomia (Word-Finding Impairment)
MeSH Terms: conditions — Aphasia; Anomia | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- anodal tDCS (Active Comparator): Intensive language therapy with anodal transcranial direct current stimulation
  Interventions: Behavioral: Intensive language therapy; Device: transcranial direct current stimulation
- sham tDCS (Sham Comparator): Intensive language therapy with Sham-tDCS
  Interventions: Behavioral: Intensive language therapy; Device: transcranial direct current stimulation

INTERVENTIONS:
Behavioral: Intensive language therapy — 2 weeks of daily computerized naming training, daily, 3 hours
Device: transcranial direct current stimulation — 1mA anodal over M1 primary motor cortex for 20min with 35cm/2 electrode, Cathode (100cm/2) contralateral

SUMMARY:
The purpose of this study is to determine if non-invasive electrical brain stimulation can enhance the outcome of intensive language therapy in chronic aphasia.

DETAILED DESCRIPTION:
Stroke is the leading cause of death and disability worldwide. Given the increasing average lifespan worldwide, the incidence and prevalence of patients with stroke will dramatically increase in the future. One of the most frequent and devastating conditions after stroke is aphasia, which affects language production and comprehension. High-frequent intensive speech-and-language therapy is currently the treatment of choice in chronic aphasia. However, despite its general effectiveness, treatment effect sizes are only low to moderate. Thus, there is a pressing need to explore novel training-adjuvant therapies to enhance treatment efficacy. Moreover, very little is known about the neurobiology of treatment-induced recovery in chronic aphasia. This is the prerequisite to improve existing and/or develop new treatment paradigms.

Thus, in the present project the investigators aim to assess whether the outcome of intensive language training can be enhanced by adjuvant non-invasive brain stimulation. They will be using anodal transcranial direct current stimulation (atDCS) that has previously been shown to enhance (a) language and motor learning in healthy subjects and (b) motor recovery in stroke patients. Specifically, in a longitudinal group comparison design, two matched groups of patients with chronic anomia will receive two weeks of intensive language training with or without atDCS. Treatment effects will be assessed immediately after the two week intervention period and several months after the end of the training. The Investigators will also use functional and structural magnetic resonance imaging (MRI) to elucidate language network changes in the two groups.

ELIGIBILITY:
Inclusion Criteria:

* chronic stroke (> 1 year after event)
* aphasia due to stroke with naming impairment
* German as first language
* first-ever stroke

Exclusion Criteria:

* more than 1 stroke
* history of severe alcohol or drug abuse, psychiatric illnesses like severe depression, poor motivational capacity
* dementia
* contraindications for Magnetic Resonance Imaging or transcranial direct current stimulation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2011-01; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
naming performance | Change of naming score from baseline (day 1 of study) to immediately after 2-week intervention period (post-testing)

SECONDARY OUTCOMES:
naming performance | Change of naming score from post-testing (after end of intervention) to 3 months after the intervention (follow-up)
Naming performance during functional magnetic resonance scanning | Change of naming score from baseline (day 1 of study) to immediately after 2-week intervention period (post-testing)
Naming performance during functional magnetic resonance imaging | Change of naming score from post-testing (after end of intervention) to 3 months after the intervention (follow-up)
Changes on the Amsterdam Nijmegen Everyday Language Test (ANELT) | Change of naming score from baseline (day 1 of study) to immediately after 2-week intervention period (post-testing)
Changes on the Amsterdam Nijmegen Everyday Language Test (ANELT) | Change of naming score from post-testing (after end of intervention) to 3 months after the intervention (follow-up)

CONTACTS AND LOCATIONS:
Overall Officials: Agnes Floeel, Prof MD, Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Charite, Berlin, Germany